CLINICAL TRIAL: NCT06327399
Title: Effect of Dexmedetomidine Infusion Dose Versus Rapid Bolus Dose on Hemodynamic Changes During Laryngoscopy and Tracheal Intubation in Adults. A Randomized Comparative Study.
Brief Title: Dexmedetomidine Infusion Dose Versus Rapid Bolus Dose Before Tracheal Intubation.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, maged gamal, Anesthesia lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS-373-2023
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Dexmedetomidine; Intubation Complication
MeSH Terms: interventions — NOP-bolus regimen; Atropine; Ephedrine; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients will receive Dexmedetomidine infusion dose of 1 mcg/kg over 10 min.
  Interventions: Drug: Dexmedetomidine infusion; Drug: Atropine Sulfate; Drug: Ephedrine; Drug: Propofol
- Group B (Active Comparator): patients will receive Dexmedetomidine bolus dose of 0.3 mcg/kg over 60 seconds.
  Interventions: Drug: Dexmedetomidine bolus; Drug: Atropine Sulfate; Drug: Ephedrine; Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine infusion — patients will receive Dexmedetomidine infusion dose of 1 mcg/kg over 10 min before induction.
  Other Names: infusion
  Arms: Group A
Drug: Dexmedetomidine bolus — patients will receive Dexmedetomidine bolus dose of 0.3 mcg/kg over 60 seconds.
  Other Names: Bolus
  Arms: Group B
Drug: Atropine Sulfate — If heart rate falls below 45 bpm, rescue dose (500 mcg) of atropine will be given.
Drug: Ephedrine — If mean blood pressure decreases below 50 mmHg, boluses of 10 mg ephedrine will be given
Drug: Propofol — Propofol 20 mg boluses till loss of contact
  Other Names: induction of anethesia

SUMMARY:
Dexmedetomidine bolus dose may provide similar or less hemodynamic changes (less bradycardia and less hypertension) than infusion dose during induction of anaesthesia and tracheal intubation.

DETAILED DESCRIPTION:
Preoperative assessment of all patients undergoing elective surgical procedures under general anaesthesia comprises history taking, clinical examination, laboratory testing (complete blood count, kidney function tests, liver function tests), electrocardiogram, and chest X-ray. The study protocol will be explained to the patients, and their consent will be obtained. The patients will be continuously monitored in the operating room for heart rate, blood pressure, and oxygen saturation (baseline values). Then a 20-gauge cannula will be inserted.

Patients will be randomly assigned into two groups: Group A will receive Dexmedetomidine infusion dose of 1 mcg/kg diluted to 100 ml normal saline infused over 10 minutes and Group B will receive Dexmedetomidine bolus dose of 0.3 mcg/kg diluted to 10 mL normal saline administered intravenously over 60 seconds. Then Patients will be induced with propofol till loss of verbal contact, followed by atracurium 0.5 mg/kg IV. After 3 minutes, tracheal intubation will be performed with an appropriate size of cuffed tracheal tube and connected to end tidal CO2 monitor. After confirmation of bilateral equal air entry, it is connected to mechanical ventilation using isoflurane 1.2% for maintaining anesthesia and keeping end tidal CO2 between 35-40 mmHg, Ringer's solution at a rate 5ml/kg/hour IV will be infused for fluid maintenance. If heart rate falls below 45 bpm, rescue dose (500 mcg) of atropine will be given. If MAP decreases below 50 mmHg, boluses of 10 mg ephedrine will be given, while escalation of MAP will be treated by boluses of 50 mg propofol.

At the end of surgery, the inhaled gas is off and the patient is reversed with neostigmine 0.05mg/kg and atropine 0.01mg/kg, then extubation is done. The two groups will be observed for changes in hemodynamic parameters i.e. heart rate (HR) and mean arterial blood pressure at preinduction period (baseline), after 1 min from dexmeditomedine taking, after induction, at intubation and 1,3,5 and 10 min after intubation. No intervention will be allowed during these 10 minutes and morphine at a dose 0.1mg/kg will be used as analgesia for surgery after 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients.
* Mallampati grade I and II.

Exclusion Criteria:

* Patient refusal.
* Morbid obesity.
* Predicted difficult airway/unanticipated difficult intubation or laryngoscopic attempt lasting greater than 15 seconds or two attempts or more.
* Patients with uncontrolled sepsis.
* Pregnancy or breast feeding.
* Patients with renal impairment i.e. SCr ≥ 1.5
* Any patient on regular intake of beta blockers or calcium channel blockers.
* CNS disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-21 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Mean blood pressure upon laryngoscopy | 1 minute
  mean blood pressure measurement (mmhg) during laryngoscopy

SECONDARY OUTCOMES:
Blood pressure & Heart rate | 1 min after dexmeditomedine, after induction, at intubation and 1,3,5 and 10 min after intubation
  Heart rate (bpm), Systolic, Diastolic and Mean arterial blood pressure (mmhg)
Propfol | induction
  total boluses dose needed for induction
Bradycardia | from start of dexmedetomidine injection before induction till 10 minutes after intubation
  Number of events : If heart rate falls below 45 bpm, rescue dose (500 mcg) of atropine will be given.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided